CLINICAL TRIAL: NCT01659450
Title: Low Energy Density Diet and Weight Loss Maintenance
Brief Title: Low Energy Dense, Weight Maintenance, Risk of Cardiovascular Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Azadbakht, Principal Investigator, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Low energy density diet; IUMS (Other: Isfahan University of Medical Sciences)
Record Dates: First submitted 2012-08-01; First posted 2012-08-07 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Body Weight Decreased
Keywords: overweight; obesity; low energy dense
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low energy dense (Experimental): Diet of the LED group contained 30%fat, 15% protein and 55% carbohydrate. Most of the consumed carbohydrates in the LED diet group were fruits, vegetables and whole grains. In addition, this group received more servings of vegetables groups daily in the form of liquid diets or some menus contain more vegetables
  Interventions: Other: low energy dense; Other: diet
- control (Experimental): In the group with a control diet, 35% of the energy was provided by fat, 15% by protein and 50% by carbohydrate
  Interventions: Other: control; Other: diet

INTERVENTIONS:
Other: low energy dense — This group received a diet appropriate with their weight in the form of low energy density diet
  Other Names: LED
  Arms: Low energy dense
Other: control — This group received a diet appropriate with their weight in the form of an usual diet regarding the energy density.
  Other Names: usual
  Arms: control
Other: diet — Calorie requirements of each subject were estimated based on resting energy expenditure (by the use of Harris-Benedict equation) and physical activity levels.
  Other Names: low energy dense; control

SUMMARY:
Investigators presumed that low energy density (LED) diet consumers will have lower risk of cardiovascular disease and are able to maintain their weight longer .

DETAILED DESCRIPTION:
Previous studies introduced different dietary interventions for weight loss maintenance. Besides the debate on low fat or low carbohydrate diets, focusing on some food groups including fruits, vegetables and low fat dairies in the diet may be helpful for weight maintenance. However, energy intake is the key factor of weight maintenance. Energy intake will decrease by reducing energy density (ED) of a diet without producing short-term calorie restriction or feeling hunger. There are several studies which showed the beneficial effects of low energy density diets on weight reduction. However, few studies discuses regarding the effects of such diets on weight maintenance.

ELIGIBILITY:
Inclusion Criteria:

* who were on weight loss diet for the last one year and additionally, they did not want to lose more weight.
* Non-pregnant, non-lactaries and non-smokers aged 40-70 years included in the present study

Exclusion Criteria:

* dietary poor compliance

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
better weight maintenance by LED | 7 months

SECONDARY OUTCOMES:
better CVD risks status by LED | 7 months

OTHER OUTCOMES:
better weight control | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Leila Azadbakht, PhD, Principal Investigator — Isfahan University of Medical Sciences

REFERENCES:
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717